CLINICAL TRIAL: NCT06202001
Title: Phase I/II Study of Irinotecan Plus Trifluridine/Tipiracil (TAS-102) in Combination With Bevacizumab as a Second-Line Therapy for Patients With Metastatic Colorectal Cancer (mCRC)
Brief Title: Irinotecan, TAS-102 Plus Bevacizumab as a Second-Line Therapy in mCRC Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC3945
Record Dates: First submitted 2024-01-02; First posted 2024-01-11 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; Trifluridine; tipiracil; trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Irinotecan, TAS-102 plus Bevacizumab arm (Experimental): This study followed a classic 3+3 design, in which patients received escalating doses of TAS-102 (20, 25, 30, or 35 mg/m2/dose, administered twice daily for days 1-5) and irinotecan (135, 150, 165, or 180 mg/m2 on day 1) with a fixed dose of bevacizumab (5 mg/kg on day 1), repeated every 14 days.
  Interventions: Drug: Irinotecan, Trifluridine/tipiracil (TAS-102) plus Bevacizumab

INTERVENTIONS:
Drug: Irinotecan, Trifluridine/tipiracil (TAS-102) plus Bevacizumab — This study followed a classic 3+3 design, in which patients received escalating doses of TAS-102 (20, 25, 30, or 35 mg/m2/dose, administered twice daily for days 1-5) and irinotecan (135, 150, 165, or 180 mg/m2 on day 1) with a fixed dose of bevacizumab (5 mg/kg on day 1), repeated every 14 days.
  Other Names: Irinotecan+TAS-102+Bevacizumab

SUMMARY:
In mCRC, response to second-line chemotherapy is limited, and few treatment options are available. It is urgent to design an optimal second-line treatment regimen to improve the response rate and prolong the survival of patients with mCRC. Several studies preliminarily demonstrated that irinotecan, TAS-102 plus bevacizumab regimen could bring promising efficacy with a tolerable safety profile for patients with mCRC as a second-line treatment. This phase I/II study was aimed to determine the recommended phase II dose (RP2D) of the combination of TAS-102, irinotecan, and bevacizumab for future clinical trials in patients with mCRC refractory to both fluoropyrimidine and oxaliplatin and to evaluate its safety and preliminary efficacy.

DETAILED DESCRIPTION:
This was a single-arm, open-label, phase I, dose-escalation study to establish the recommended phase II dose (RP2D) for the combination of TAS-102, irinotecan, and bevacizumab and evaluate its safety.

This study followed a classic 3+3 design, in which patients received escalating doses of TAS-102 (20, 25, 30, or 35 mg/m2/dose, administered twice daily for days 1-5) and irinotecan (135, 150, 165, or 180 mg/m2 on day 1) with a fixed dose of bevacizumab (5 mg/kg on day 1), repeated every 14 days. Initially, three patients will receive therapy at dose level 1. If dose-limiting toxicity (DLT) occurred, an additional three patients were enrolled at the same dose level. If none of the first three patients or less than two of the six patients exhibited DLT, then the study regimen was escalated to a higher dose level. If two or more DLTs occurred, the study regimen was reduced to a lower dose level.

The maximum tolerated dose (MTD) was defined as the highest dose level at which less than one-third of evaluable patients treated had a DLT during the first or second cycle of drug administration. The RP2D was defined as the MTD. At least six patients at the MTD or RP2D were needed to estimate these doses accurately.

Treatment was continued until RECIST-defined disease progression or clinical disease progression, unacceptable toxicity, patient request to withdraw treatment, and a treatment-free period of >30 consecutive days.

Adverse events (AEs) were graded based on the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.

The response was assessed by the investigator according to RECIST version 1.1.

ELIGIBILITY:
Inclusion Criteria:

1. Colorectal adenocarcinoma confirmed histologically or histopathologically.
2. Patients were clinically diagnosed with metastatic colorectal cancer based on computed tomography (CT) scan and magnetic resonance imaging (MRI) according to AJCC 8th edition.
3. Patients have received oxaliplatin-based first-line chemotherapy with or without targeted therapy, immunotherapy or radiotherapy.
4. Age ≥18 and ≤70.
5. ECOG physical status score is 0 or 1, and no obvious deterioration within 2 weeks prior to use on Day 1 of Cycle 1.
6. Appropriate organ function according to the following laboratory test values:

   1. Hemoglobin value ≥90g/L.
   2. White blood cell count ≥3.5*109/L.
   3. Absolute neutrophil count ≥1.5*109/L.
   4. Platelet count ≥100*109/L.
   5. Serum creatinine ≤ upper limit of normal (ULN) or creatinine clearance ≥60ml/min.
   6. Total serum bilirubin ≤1.5* upper normal limit (ULN).
   7. Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤2.5* upper limit of normal value (ULN).
7. Signed the informed consent.

Exclusion Criteria:

1. The pathological types were squamous carcinoma, neuroendocrine carcinoma, adenosquamous carcinoma, and other histological types except adenocarcinoma.
2. Patients who had shown hypersensitivity to Irinotecan and Trifluridine/tipiracil (TAS-102) or any other component of them. Patients who previously received irinotecan while disease progressed. However, patients who previously received irinotecan while progressing during maintenance therapy are eligible.
3. Known hypersensitivity to Bevacizumab or hypersensitivity to any other component of Bevacizumab.
4. Patients unable to swallow or lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome, or inability to take oral medication.
5. Patients had recurrent episodes of bleeding (risk of gastrointestinal bleeding) or received transfusions in the previous 2 weeks.
6. Major surgery in the previous 4 weeks. (Biopsy is excluded)
7. Previous or concurrent cancer diagnosed within 5 years prior to study inclusion, except for curatively treated in situ cervical cancer, non-melanoma skin cancer, basal cell carcinoma, benign prostate cancer, ductal carcinoma in situ, well-differentiated thyroid cancers and superficial bladder tumors: staged Ta (non-invasive tumor), Tis (carcinoma in situ), and T1 (tumor with lamina propria invasion). Carcinomas that can be cured by adequate treatment are also excluded.
8. History of abdominal fistula, gastro-intestinal perforation, intestinal obstruction, chronic diarrhea or inflammatory bowel disease including Crohns disease and ulcerative colitis within 6 months prior to the first study treatment.
9. Patients with severe cardiac dysfunction, such as LVEF< 50%, CHF≥ grade 2, severe/unstable angina, history of stroke or transient ischemic attack or myocardial infarction in the previous 6 months.
10. Uncontrolled hypertension (systolic blood pressure >160 mmHg or diastolic pressure >100 mmHg despite treatment) and uncontrolled diabetes (fasting plasma glucose > 8.9 mmol/l).
11. Patients with a history of ventricular tachycardia, torsades de pointes, prolonged QTc, complete left bundle branch block or third-degree atrioventricular conduction block.
12. Patients with active hepatitis B, hepatitis C, syphilis or human immunodeficiency virus infection.
13. Arterial or venous thrombotic or embolic events such as deep vein thrombosis, and pulmonary embolism within 3 months of starting study treatment (catheter-related thrombosis is excluded).
14. Patients with active pulmonary tuberculosis were taking anti-tuberculosis treatment or have taken anti-tuberculosis treatment within 12 months of starting study treatment.
15. Patients with severe primary respiratory diseases, interstitial lung disease, or history of pneumonitis.
16. Patients with current active infections requiring anti-infection treatment within 2 weeks of starting study treatment.
17. Patients with a history of psychiatric drug abuse or a history of drug abuse.
18. Pregnant or lactating women.
19. Patients of childbearing potential are unwilling to practice contraception.
20. Patients with any clinically significant disease, metabolic disorders or laboratory abnormality. Investigator could reasonably consider those patients not suitable for the study, affecting the results analysis or putting those patients at high risk.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 36 months
  The proportion of patients with a confirmed complete response or partial response using RECIST 1.1

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 36 months
  The time from the date of the first administration of this regimen to the date of first documented disease progression or death due to any cause
Overall Survival (OS) | 36 months
  The time from the initiation of the first dose of medication in a patient to death from any cause.
Safety and tolerability by incidence, severity and outcome of adverse events | 36 months
  Safety and tolerance will be evaluated by incidence, severity and outcomes of adverse events (AEs) and categorized by severity in accordance with the NCI CTC AE Version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Yongkun Sun, Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China